CLINICAL TRIAL: NCT04090216
Title: In-Hospital Outcome of Primary Percutaneous Coronary Intervention in Addict ST Elevation Myocardial Infarction Patients in Assuit University Hospital.
Brief Title: Outcome of Primary PCI in STEMI Addict Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdalla Aly, Abdalla Aly Gamal, Assiut University
Other Study IDs: Primary PCI
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Addict patients: patients with substance use disorders presented with STEMI & undergoing Primary PCI
  Interventions: Device: Primary Percutaneous Coronary Intervention
- Non Addict patients: patients without substance use disorders presented with STEMI & undergoing Primary PCI
  Interventions: Device: Primary Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Primary Percutaneous Coronary Intervention — Primary PCI will be done for patients with STEMI in both groups of patients

SUMMARY:
• The goal of this study is to Identify the in-hospital outcome of primary PCI in treatment of STEMI in addict patients in comparison to non-addict patients.

DETAILED DESCRIPTION:
Myocardial infarction (MI), is a type of acute coronary syndrome, in which there is damage to the cardiac muscle as demonstrated by increased cardiac Troponin levels in the setting of acute ischemia (1). Myocardial infarction (MI) is a fatal disease that is caused by block in the oxygen supply of blood vessels of the heart muscle, leading to permanent heart muscle damage and death of its cells. According to world health organization (WHO) report published in 2014, 68% of global deaths annually related to non communicable diseases, Cardiovascular diseases constitute 31% of these deaths denoting that they are the leading cause of death (2). Risk factors of cardiovascular diseases include behavioral factors as eating un healthy food, smoking, alcohol intake, and other substance abuse.

Regarding management of MI, There have been several studies that have shown the superiority of percutaneous coronary intervention (PCI) as a treatment for ST-elevation myocardial infarction (STEMI) when compared with thrombolytic therapy in terms of reducing mortality rate and recurrence of myocardial infarction (MI) [3-5].

Regarding Drug abuse cardiovascular effects. It depends on the drug, dose, and route of administration, cardiovascular consequences can range from innocuous side effects, to life threatening ventricular arrhythmias and myocardial infarction.

Sympathomimetic drugs like amphetamines cause an increase in release of peripheral catecholamines stimulating increases in heart rate, systemic vascular resistance, and cardiac contractility, thus resulting in augmentation of cardiac output and blood pressure. In contrast, several drugs are directly cardiodepressant in the acute setting, and many drugs of both types are cardiotoxic causing cardiomyopathy and congestive heart failure with long-term use.

Changes in the balance of myocardial oxygen supply and demand with drug use can lead to myocardial ischemia. For example, cocaine increases oxygen demand in the myocardium while simultaneously decreasing supply by inducing epicardial coronary vasoconstriction. Modulation of lipid profiles, coagulation factors, platelet function, and inflammation further heighten the risk of cardiac ischemic events in patients using these drugs.

Many recreational drugs are arrhythmogenic in the acute setting or during abstinence/withdrawal. Mechanisms of arrhythmias are complex and likely result from interplay between the direct effects of drugs, electrolyte derangements, sympathetic nervous alterations, and cardiac ischemia.(6)

Substance Use Disorders (SUD) are considered to be prevalent In Middle Eastern Arab countries, particularly Egypt, but there is scarce information on the problem of patients with substance abuse or dependence attending emergency rooms in general hospitals.

In across sectional study done in EL Mansoura University in 2012, Among patients with substance abuse, cannabis ranked first (3.6%) then tramadol 1.8%, polysubstance1.7%, followed by stimulants group (1.3%), alcohol (1.1%), and finally anticholinergics (0.5%) and volatile substances (0.3%). Urine toxicology shows that 30% used at least one of these illicit drugs: (20%) tested positive for cannabis, (6%) had a positive urine screen for amphetamine, and (10%) tested positive for opiates.(7)

Prior studies have reported discrepant results on the association between substance use disorders and access to Primary PCI after acute myocardial infarct (AMI) [8]. Druss and colleagues showed that patients with SUDs aged 65 and older in acute care non-governmental hospitals in the United States were less likely than those with neither mental nor substance use disorder to receive cardiac catheterization after acute MI [9]. Young reported data stratified by age, indicating that patients with SUDs both younger and older than 65 years have lower rates of cardiac procedures and higher rates of in-hospital mortality compared with those with neither mental nor substance use disorders [10]. Most recently, Jones and colleagues published results from an analysis of administrative data from a large commercially insured sample of all ages, adjusting for comorbidities.(11) They obtained an unexpected result: those with SUDs were more likely to receive percutaneous coronary intervention (PCI) in comparison to those with neither mental nor substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* All patients of all categories of ages who will be presented with ST elevation myocardial infarction and undergoing primary PCI in Assuit University Hospital.

Exclusion Criteria:

* -Patients who present with STEMI but will not undergo primary PCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: : The study will include all patients presented with ST elevation myocardial infarction undergoing primary PCI in Assuit University Hospital , Patients will be classified into 2 groups : Group A:patients proved to be addicts by DSM-5 criteria of WHO for addiction & urine tests.
  Group B: Non-addict patients .
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
outcome of primary PCI in addict STEMI patients | 30 minutes
  Identify the in-hospital outcome of primary PCI in treatment of STEMI in addict patients in comparison to non-addict patients.

REFERENCES:
- See also: .World Health Organization (2014): Global status report on noncommunicable diseases. https://en.wikipedia.org/wiki/World_Health_Organization — http://en.wikipedia.org/wiki/World_Health_Organization